CLINICAL TRIAL: NCT00004816
Title: A Maintenance Extension of Phase I Pilot Study of Chimeric Anti-CD4 Antibody M-T412 in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Stanford University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 199/12050; SUMC-C0128T03
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Multiple Sclerosis; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Drug: monoclonal antibody M-T412

SUMMARY:
OBJECTIVES: I. Evaluate the safety and immunogenicity of single and multiple doses of M-T412, a chimeric murine-human anti-CD4 monoclonal antibody, in patients with multiple sclerosis.

II. Evaluate the pharmacokinetics of M-T412. III. Obtain preliminary data on the clinical response to M-T412.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is an open label, dose escalating study. Escalating doses of M-T412 are administered to cohorts of 5 patients each receiving a single dose intravenously over 2 hours.

Patients who complete the single dose assessment of M-T412 may receive up to 3 additional single doses of M-T412 IV over 2 hours, with each repeated dose given at least 1 month apart.

Then, patients receive one dose level of M-T412 IV over 2 hours at 3 month intervals over a period of 12 months for a total of 5 doses. Once recovery of CD4 cells is obtained, the next scheduled infusion of M-T412 begins. Patients are omitted from study if CD4 cells remain attenuated following 2 scheduled infusion sessions.

Patients are followed at 3, 6, 12, and 24 months after the first infusion.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of chronic, advanced, progressive multiple sclerosis (MS)

--Prior/Concurrent Therapy--

* Biologic therapy: No sensitivity to murine proteins No prior treatment at any time with anti-CD4 antibodies, other murine antibodies, or other anti-T cell antibodies (e.g., xenologous or human) At least 4 weeks since use of other biological agents
* Chemotherapy: No concomitant chemotherapy At least 3 months since prior chemotherapy
* Endocrine therapy: No concomitant steroidal therapy At least 3 months since prior steroidal therapy
* Radiotherapy: No total lymphoid irradiation prior to study No concomitant radiotherapy At least 3 months since prior radiotherapy
* Other: No use of investigational drugs within 30 days prior to study

--Patient Characteristics--

* Age: 21 to 75
* Hematopoietic: Hemoglobin at least 10 g/dL WBC at least 4000/mm3 Granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 CD4+ lymphocyte count at least 300 cells/mm3
* Other: Not pregnant or lactating Effective contraception required of fertile patients for 3 months prior to and during study No substance abuse (e.g., drug or alcohol) Not HIV positive No AIDS-Related Complex (ARC) No serum antibodies to HIV Negative serum antibody test for HIV within 1 month prior to study No underlying medical or psychiatric condition

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 1995-07

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Steinman, Study Chair — Stanford University